CLINICAL TRIAL: NCT03643926
Title: Arthroscopic Versus Open Brostrom for Ankle Instability: a Randomized Clinical Trial
Brief Title: Arthroscopic Versus Open Brostrom for Ankle Instability
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Nacime Salomão Barbachan Mansur, Principal Investigator, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13072018
Record Dates: First submitted 2018-08-15; First posted 2018-08-23 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Ankle Sprains; Instability, Joint; Ligament Injury; Surgery
Keywords: ankle; instability; brostrom; open; arthroscopic
MeSH Terms: conditions — Ankle Injuries; Joint Instability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arthroscopic Brostrom (Experimental)
  Interventions: Procedure: Arthroscopic Brostrom
- Open Brostrom (Active Comparator)
  Interventions: Procedure: Open Brostrom

INTERVENTIONS:
Procedure: Arthroscopic Brostrom — Brostrom-Gould lateral ligament ankle reconstruction performed by arthroscopic view
  Arms: Arthroscopic Brostrom
Procedure: Open Brostrom — Brostrom-Gould lateral ligament ankle reconstruction performed by an open approach.
  Arms: Open Brostrom

SUMMARY:
Background: Ankle sprains are among the most prevalent lesions in primary care. A substantial number of these ligament lesions will develop ankle instability and require a surgical procedure. The Brostrom-Gould technique is the standard surgical approach for this condition, providing excellent results over the years. Thru the last decades, the arthroscopic Brostrom has gain popularity and support by several studies. Yet, there is no consensus regarding the best procedure to treat ankle instability nowadays.

Hypothesis: The arthroscopic Brostrom technique will present better levels of pain and function when compared to the standard open approach.

Design: blinded, in parallel groups, multicentric, randomized, clinical trial.

Materials and Methods: 98 patients with a diagnosis of chronic ankle instability, referred from primary or secondary health care services, will be assessed and enrolled in this study. Participants will be divided in two groups (randomized by sequentially numbered identical envelopes, which will be administered serially to participants), one containing the open Brostrom repair technique and the other comprehending the arthroscopic Brostrom approach. The assessments will occur in 3, 6, 12, 24 and 48 weeks. Patients will be evaluated primarily by complications and secondarily the Cumberland Ankle Instability Tool (CAIT), American Orthopedic Foot and Ankle Society (AOFAS), the Visual Analogue Scale (VAS), the Foot Function Index (FFI) and the 36 Item Short Form Health Survey (SF-36). The investigators will use Comparison of Two Proportions via relative frequency analysis, the Pearson Correlation the Chi-Square test and the ANOVA for statistical analyses.

Discussion: This study intends to establish if the arthroscopic Brostrom technique can produce excellent and reliable results when treating chronic ankle instability. A shorter surgical time, a better cosmetic appearance and a smaller soft tissue injury would support the choice for this procedure if the outcomes could be compared to the open approach.

DETAILED DESCRIPTION:
1. Introduction

   Ankle sprains are among the most prevalent lesions in the athletic and non-athletic population(1). Accounting to up than 14% of emergency visits and with an estimated year cost of more than U$6 billion, it has a high impact in the health care system(2,3). Approximately 10 to 40% of these cases will develop ankle instability. The most susceptive population are those with an erratic treatment and/or poor rehabilitation program(4). Over the past years, the open Brostrom Gould procedure has been state as the gold standard procedure for this specific group of patients. (5,6). (7,8).

   With the development and improvement intra-articular ligament reconstruction and repair for shoulder and knee, the possibility to perform the same type of procedure at the ankle has grown. Arthroscopic-assisted Brostrom techniques were first described by Nery et al and Corte-Real et al near the year 2010(9,10). Some authors proposed modifications to these original approaches, but the main surgery concept was maintained(11-14).. During the last few years, a good number of studies were able to present good clinical and functional results with this procedure(1,11,15-18).

   Ankle arthroscopy is a reliable procedure and has been indicated to evaluate and treat a great number of ankle pathologies over the past decades(19,20). Ankle impingement, osteochondral lesions and tibiotarsi arthrodesis are some of the conditions that have good literature support in favor for the arthroscopic approach(21). Also, its use, prior to an ankle ligament repair or reconstruction, is advocated and sustained by several studies(22-26). It allows a complete articular visualization, providing the surgeon with a definitive scenario when dealing with ankle instability. Cartilage lesions, impingement syndromes and loose bodies that could be neglected by subsidiary exams can be detected and treated arthroscopically.

   The intra-articular ligament reconstruction and repair is not novelty for others orthopedic areas. The development of the anterior cruciate ligament surgery went to from the open approach to the arthroscopic technique over the last decades until the least was proclaimed the gold standard(27,28). The Bankart lesion, a condition normally related to traumatic shoulder instability, has a similar history, although the arthroscopic approach wasn't able to produce superior general results when compared to its open counterpart (29,30). Advances in the "all-inside" ligament repair are taking place at the shoulder and hip segment as well, showing promising and solid outcomes(31,32).

   Despite all the solid results regarding the biomechanical profile and the clinical effects of the arthroscopic Brostrom, there is a gap in its bibliography when it comes to high-level studies. Only Yeo et al in 2016 were able to show similar results between the open and the all-inside procedures with one-year follow-up study (1). Lately, an attempt in producing on systematic review on the subject was published, but no clinical trials were found to be included(33).

   Herein, our objective is to evaluate the effectiveness of the arthroscopic Brostrom technique and compare it to the open Brostrom procedure regarding complications, function by the Cumberland Ankle Instability Tool (CAIT), the American Orthopedic Foot and Ankle Society score (AOFAS), the Foot Function Index (FFI) and the 36 Short Form Survey (SF-36). The primary hypothesis is that the arthroscopic Brostrom will mitigate pain and improve function as compared to the open approach.
2. Material and Method

2.1 Design, setting and recruitment

This will be a multicentric, with parallel groups, randomized clinical trial. The study will be conducted at São Paulo Hospital, a tertiary, teaching hospital fully affiliated with the Federal university of São Paulo (UNIFESP), and at Hospital das Clínicas, another tertiary, teaching hospital fully affiliated with the Federal university of Minas Gerais (UFMG).

Participants will be enrolled at both hospitals, which provide assessment and treatment to approximately 5 (five) new patients with ankle instability per week. They will be referred by local orthopedist doctors or health professionals. The information to these physicians will be delivered by e-mail addressed directly to them, as well as via posters exhibited in places containing orthopedic medical care (outpatient clinic, emergency room).

2.2 Inclusion Criteria

* Individuals must be older than 18 and younger than 65 years of age, both genders;
* Participants must be experiencing instability symptoms at the ankle over the last six months;
* Clinical diagnosis of ankle instability, defined as the presence of at least one previous ankle sprain associated with a current instability sensation by the patient and the presence of a positive anterior drawer test; the previous lateral ligament injury must be confirmed by Magnetic Resonance Imaging (MRI) findings.

2.3 Exclusion Criteria

* Previous surgery involving the affected foot or ankle;
* History or documented evidence of autoimmune or peripheral vascular diseases;
* History or documented evidence of peripheral neuropathy (nervous compression syndrome, tarsal tunnel syndrome) or systemic inflammatory disease a (rheumatoid arthritis, spondylitis, Reiter Syndrome, etc.);
* Associated injuries, such as osteochondral lesions, tendon ruptures and fractures;
* Associated instability, such as syndesmotic and medial instability;
* Cavovarus foot;
* BMI over 35;
* Previous infiltration in the ankle over the six months preceding the initial assessment;
* Pregnancy;
* Any condition that represents a contraindication of the proposed therapies;
* Impossibility or incapacity to sign the informed Consent Form;
* History or documented evidence of blood coagulation disorders (including treatment with anti-coagulants, but excluding aspirin);
* Use of heart pacemaker;
* Presence of infectious process (superficial on skin and cellular tissue, or deep in the bone) in the region to be treated;

2.4 Sampling

The objective of this study is to right evaluate the efficacy of the Brostrom arthroscopic technique and compare it to the open Brostrom procedure in relation to the function by the American Orthopedic Foot and Ankle Society Score (AOFAS), the foot function Index (FFI) and o 36 Short Form Survey (SF-36).

Thus, considering a 7.2 million population in the city of Sao Paulo that fit the criteria of inclusion and/or exclusion (Source: Census 2010) and respecting an involvement index of 0.072% value (0.72 by 1000 Exposition, according to the Ankle Consortium). Therefore, the target population estimated for the study is 5,155 people.

Using the formula shown in appendix I to calculate the sample size with a 10% error, we estimated a sampling of 98. This sample quantity was defined according to the methodology expressed in appendix I, where, based in the central boundary theorem and the laws of large numbers, this sample size ensures that statistical analyses will be reliable.

2.5 Procedures

A written, signed and dated informed consent will be obtained from the subject before any study-related procedures are performed. The patients will have to fill out an initial questionnaire in order to be enrolled (Attachment 2). After that, the assistant doctor will do the physical diagnostic examination. Then, X-rays and the MRI procedures will take place, to complete the diagnostic assessment. The patient will be included in the protocol and duly randomized after the diagnostic confirmation and fulfilment of all the inclusion criteria and non-adequacy to the exclusion criteria.

The randomization sequence will be generated via computing software (http://www.randomizer.org/form.htm), producing a list from 1 - 98, and each number will be related to a sole treatment method. We will do a randomization with interchanged blocks, with the same number of patients in each group.

Each non-transparent, opaque, sealed envelope, numbered from 1 to 98, will contain either a paper with the word "open" or with the words "arthroscopic". Each treatment method will have the same number of envelopes. The patients will be initially assessed individually, being randomized and allocated in the same way. The intervention procedures will be the same, with the same positioning and preparations, but differing regarding the lateral ligament repair approach.

The evaluator doctor won't have access to the protocol test applied to each patient, and the surgeries (open or arthroscopic) will be conducted by different physicians. The patients in both groups will receive a large bandage at the operation site before every consultation, blinding the evaluator.

2.6 Interventions 2.6.1 Open Brostrom Approach

1. Period from diagnosis to intervention: up to 1 month.
2. Patient will receive a general anesthesia and a popliteal peripheral block. After surgical site preparation, the traditional arthroscopic portals will be performed.
3. An ankle arthroscopy will be held, to confirm the nonexistence of chondral lesions, medial instability or syndesmotic instability. The ankle will be cleaned, and all impingements removed. The proximal ligament insertion at the lateral malleolus will be debrided.
4. All the arthroscopic instruments will be removed. A lateral longitudinal incision will be held over the lateral capsule. The fibula apex, at the ATFL and CFL footprint, will receive a 3.0mm suture anchor (with two n2 high-resistant sutures).
5. The ligaments will be reattached with tension in a paints-over-vest fashion, using one suture for the ATFL region and one for the CFL region.
6. The incisions will be closed, and the patient placed in a post-operative boot. Weight-bearing will start at the 1st week (with the boot) and range of motion (ROM) will begin at the 3rd week (limiting inversion until the 6th week). Patients will be transitioned to an ankle brace at the 4th week.
7. Patients will be evaluated, and the questionnaires applied at the 3rd, 6th, 12th, 24th and 48th post-operative week.

2.6.2 Arthroscopic Brostrom Approach

1. Period from diagnosis to intervention: up to 1 month.
2. Patient will receive a general anesthesia and a popliteal peripheral block. After surgical site preparation, the traditional arthroscopic portals will be performed.
3. An ankle arthroscopy will be held, to confirm the nonexistence of chondral lesions, medial instability or syndesmotic instability. The ankle will be cleaned, and all impingements removed. The proximal ligament insertion at the lateral malleolus will be debrided.
4. The fibula apex (by arthroscopic view), at the ATFL and CFL footprint, will receive a 3.0mm suture anchor (with two n2 high-resistant sutures).
5. One suture will be passed at the most superior anterolateral capsular site and the other at the most inferolateral capsular site, respecting the safe zone between the superficial fibular nerve and the peroneal tendons. These maneuvers will be executed in a percutaneous and arthroscopic assisted technique. The ligaments will be reattached with tension using an arthroscopic knot.
6. The incisions will be closed, and the patient placed in a post-operative boot. Weight-bearing will start at the 1st week (with the boot) and range of motion (ROM) will begin at the 3rd week (limiting inversion until the 6th week). Patients will be transitioned to an ankle brace at the 4th week.
7. Patient will be evaluated, and the questionnaires applied at the 3rd, 6th, 12th, 24th and 48th post-operative week.

2.6.3 Adjuvant therapies

Both groups will be submitted to the same post intervention care program, and they will be advised to use the following adjuvant therapies according to the intensity of their symptoms:

Elevation Every patient will be oriented to perform limb elevation during the post-operative period.

Pain Killers

Level 1:

* Dipyrone 1g every 6 hours, in case of pain, or
* Paracetamol 750mg every 6 hours

Level 2 (in case the pain does not diminish with level 1):

* Tramadol 50mg every 6 hours, in case of pain, or
* Codeine 30mg every 6 hours, in case of pain. The patient must present, at each visit to the doctor, the daily annotation concerning the used sedative medication. The medication will be supplied to the patient after the intervention, with the respective orientation concerning its use. After the period of five days of sedation, in case the pain persists, the patient will be reassessed, to check the necessity of changing the medication. If after the sixth week assessment the pain is stronger than in the initial painful stage, the patient will have the option of either change the treatment or being excluded from the study.

2.7 Primary outcome

• Major complications such as dehiscence, neural damage, infection and re-rupture.

Significant difference between groups.

* Dehiscence: inability to heal the soft tissue coverage until the end of the 4th post-operative week.
* Peripherical nerve damage: hypoesthesia or paresthesia not solved until the end of the 6th month after the surgery.
* Infection: clinical signs infection or pus drainage at the wound that required the use of antibiotics.
* Re-rupture: an ankle sprain event during the follow-up.

2.8 Secondary outcomes

* CAIT
* VAS
* FFI
* AOFAS score
* SF-36
* Minor complications such as neuropraxia and prominent suture knots.

2.9 Subject Discontinuation

Subjects may be discontinued from the study at any time. Reasons for discontinuation include:

1. Voluntary discontinuation by the subject without prejudice to further treatment.
2. Development of Complex Regional Pain Syndrome or any huge inflammatory response.
3. Pain and function severe impairment.

2.10 Statistical Analysis: After collecting the information, we will characterize the relative frequency (percentages) distribution of the qualitative variables through the Equal Test of Two Proportions. For relationship between qualitative variables analysis, the Chi-Squared test will be used. If a correlation between quantitative covariables reveals necessary, the Pearson's Correlation Test will be used. For the quantitative covariant comparison (effect measurement), we will make use of the ANOVA test.

3. Discussion Chronic ankle instability (CAI) can be a consequence in up to 40% of ankle sprains. Considering that this type of trauma can occur in more than 10,000 Americans per day and consume more than U$6 billion in related costs per year, it's fair to say that we might be dealing with a worldwide public health challenge. Although this instability may be managed with conservative treatment, many patients will require surgical resolution due their demands and expectations.

In this scenario, the Brostrom-Gould technique has emerged as the standard procedure in ankle instability operative care. Based on sustained and long-term results, its open fashion still is the preferable procedure for most of the Foot and Ankle and Sports Traumatology surgeons. Meanwhile, orthopedic arthroscopic techniques have progressed over the past decades and at the end of this century's first decade, the all-inside ankle ligament reconstruction started to be performed and published.

A moderate number of surveys regarding these techniques in the past few years showed its efficacy and safety. Yet, there is no consensus concerning what is the best way to approach ankle instability when contrasting the open and the arthroscopic approach due the lack of quality comparative studies. Our research intends to try to answer this question by a randomized clinical trial with robust outcomes and a long follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Individuals must be older than 18 and younger than 65 years of age, both genders;
* Participants must be experiencing instability symptoms at the ankle over the last six months;
* Clinical diagnosis of ankle instability, defined as the presence of at least one previous ankle sprain associated with a current instability sensation by the patient and the presence of a positive anterior drawer test; the previous lateral ligament injury must be confirmed by Magnetic Resonance Imaging (MRI) findings.

Exclusion Criteria:

* Previous surgery involving the affected foot or ankle;
* History or documented evidence of autoimmune or peripheral vascular diseases;
* History or documented evidence of peripheral neuropathy (nervous compression syndrome, tarsal tunnel syndrome) or systemic inflammatory disease a (rheumatoid arthritis, spondylitis, Reiter Syndrome, etc.);
* Associated injuries, such as osteochondral lesions, tendon ruptures and fractures.
* Associated instability, such as syndesmotic and medial instability.
* Cavovarus foot;
* BMI over 35;
* Previous infiltration in the ankle over the six months preceding the initial assessment;
* Pregnancy;
* Any condition that represents a contraindication of the proposed therapies;
* Impossibility or incapacity to sign the informed Consent Form;
* History or documented evidence of blood coagulation disorders (including treatment with anti-coagulants, but excluding aspirin);
* Use of heart pacemaker;
* Presence of infectious process (superficial on skin and cellular tissue, or deep in the bone) in the region to be treated;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-05 (Estimated)

PRIMARY OUTCOMES:
Complications (change) | 3, 6, 12, 24 and 48 weeks
  * Dehiscence: inability to heal the soft tissue coverage until the end of the 4th post-operative week.
  * Peripherical nerve damage: hypoesthesia or paresthesia not solved until the end of the 6th month after the surgery.
  * Infection: clinical signs of site infection or pus drainage at the wound that required the use of antibiotics.
  * Re-rupture: an ankle sprain event during the follow-up.

SECONDARY OUTCOMES:
Cumberland Ankle Instability Tool - CAIT (change) | 3, 6, 12, 24 and 48 weeks
  Ankle Instability Measurement (0 to 30; higher = better)
American Orthopedic Foot and Ankle Society - AOFAS (change) | 3, 6, 12, 24 and 48 weeks
  AOFAS Hindfoot Scale for Function (0 to 100; higher = better)
Visual Analogue Scale - VAS (change) | 3, 6, 12, 24 and 48 weeks
  Pain assessment (0 to 10; higher = worse)
Foot Function Index - FFI (change) | 3, 6, 12, 24 and 48 weeks
  Global Foot Function (0 to 100%; higher = worse)
36 Item Short Form Health Survey - SF36 (change) | 3, 6, 12, 24 and 48 weeks
  Quality of Life (0 to 100%; higher = better)
Minor complications (change) | 3, 6, 12, 24 and 48 weeks
  Such as neuropraxia and prominent suture knots

CONTACTS AND LOCATIONS:
Overall Officials: Marcel JS Tamaoki, PhD, Study Chair — Federal University Sao Paulo; Caio Nery, PhD, Study Director — Federal University Sao Paulo; Fabio Matsunaga, PhD, Study Director — Federal University Sao Paulo; Roberto Zambelli, MD, Study Director — Federal University of Minas Gerais
Locations (2):
- Brazil (2):
  - Federal University of Minas Gerais, Belo Horizonte, Minas Gerais
  - Federal University of Sao Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
We intend to share all the IPD available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After statistical analysis closure.
Access Criteria: Registered researches that request access.

REFERENCES:
- [Background] Yeo ED, Lee KT, Sung IH, Lee SG, Lee YK. Comparison of All-Inside Arthroscopic and Open Techniques for the Modified Brostrom Procedure for Ankle Instability. Foot Ankle Int. 2016 Oct;37(10):1037-1045. doi: 10.1177/1071100716666508. Epub 2016 Sep 13. PMID 27623732
- [Background] McGovern RP, Martin RL. Managing ankle ligament sprains and tears: current opinion. Open Access J Sports Med. 2016 Mar 2;7:33-42. doi: 10.2147/OAJSM.S72334. eCollection 2016. PMID 27042147
- [Background] Gribble PA, Bleakley CM, Caulfield BM, Docherty CL, Fourchet F, Fong DT, Hertel J, Hiller CE, Kaminski TW, McKeon PO, Refshauge KM, Verhagen EA, Vicenzino BT, Wikstrom EA, Delahunt E. 2016 consensus statement of the International Ankle Consortium: prevalence, impact and long-term consequences of lateral ankle sprains. Br J Sports Med. 2016 Dec;50(24):1493-1495. doi: 10.1136/bjsports-2016-096188. Epub 2016 Jun 3. PMID 27259750
- [Background] Doherty C, Bleakley C, Hertel J, Caulfield B, Ryan J, Delahunt E. Recovery From a First-Time Lateral Ankle Sprain and the Predictors of Chronic Ankle Instability: A Prospective Cohort Analysis. Am J Sports Med. 2016 Apr;44(4):995-1003. doi: 10.1177/0363546516628870. Epub 2016 Feb 24. PMID 26912285
- [Background] Hamilton WG, Thompson FM, Snow SW. The modified Brostrom procedure for lateral ankle instability. Foot Ankle. 1993 Jan;14(1):1-7. doi: 10.1177/107110079301400101. PMID 8425724
- [Background] Karlsson J, Bergsten T, Lansinger O, Peterson L. Surgical treatment of chronic lateral instability of the ankle joint. A new procedure. Am J Sports Med. 1989 Mar-Apr;17(2):268-73; discussion 273-4. doi: 10.1177/036354658901700220. PMID 2667383
- [Background] Messer TM, Cummins CA, Ahn J, Kelikian AS. Outcome of the modified Brostrom procedure for chronic lateral ankle instability using suture anchors. Foot Ankle Int. 2000 Dec;21(12):996-1003. doi: 10.1177/107110070002101203. PMID 11139039
- [Background] Paden MH, Stone PA, McGarry JJ. Modified Brostrom lateral ankle stabilization utilizing an implantable anchoring system. J Foot Ankle Surg. 1994 Nov-Dec;33(6):617-22. PMID 7894411
- [Background] Nery C, Raduan F, Del Buono A, Asaumi ID, Cohen M, Maffulli N. Arthroscopic-assisted Brostrom-Gould for chronic ankle instability: a long-term follow-up. Am J Sports Med. 2011 Nov;39(11):2381-8. doi: 10.1177/0363546511416069. Epub 2011 Jul 29. PMID 21803979
- [Background] Corte-Real NM, Moreira RM. Arthroscopic repair of chronic lateral ankle instability. Foot Ankle Int. 2009 Mar;30(3):213-7. doi: 10.3113/FAI.2009.0213. PMID 19321097
- [Background] Cottom JM, Rigby RB. The "all inside" arthroscopic Brostrom procedure: a prospective study of 40 consecutive patients. J Foot Ankle Surg. 2013 Sep-Oct;52(5):568-74. doi: 10.1053/j.jfas.2013.02.022. Epub 2013 May 11. PMID 23669003
- [Background] Matsui K, Takao M, Miyamoto W, Innami K, Matsushita T. Arthroscopic Brostrom repair with Gould augmentation via an accessory anterolateral port for lateral instability of the ankle. Arch Orthop Trauma Surg. 2014 Oct;134(10):1461-7. doi: 10.1007/s00402-014-2049-x. Epub 2014 Jul 12. PMID 25015792
- [Background] Molloy AP, Ajis A, Kazi H. The modified Brostrom-Gould procedure--early results using a newly described surgical technique. Foot Ankle Surg. 2014 Sep;20(3):224-8. doi: 10.1016/j.fas.2014.01.002. Epub 2014 Jan 30. PMID 25103713
- [Background] Acevedo JI, Mangone P. Arthroscopic brostrom technique. Foot Ankle Int. 2015 Apr;36(4):465-73. doi: 10.1177/1071100715576107. Epub 2015 Mar 5. PMID 25743426
- [Background] Maffulli N, Del Buono A, Maffulli GD, Oliva F, Testa V, Capasso G, Denaro V. Isolated anterior talofibular ligament Brostrom repair for chronic lateral ankle instability: 9-year follow-up. Am J Sports Med. 2013 Apr;41(4):858-64. doi: 10.1177/0363546512474967. Epub 2013 Feb 6. PMID 23388673
- [Background] Li HY, Zheng JJ, Zhang J, Cai YH, Hua YH, Chen SY. The improvement of postural control in patients with mechanical ankle instability after lateral ankle ligaments reconstruction. Knee Surg Sports Traumatol Arthrosc. 2016 Apr;24(4):1081-5. doi: 10.1007/s00167-015-3660-2. Epub 2015 May 28. PMID 26017745
- [Background] Nery C, Fonseca L, Raduan F, Moreno M, Baumfeld D; ESSKA AFAS Ankle Instability Group. Prospective study of the " Inside-Out" arthroscopic ankle ligament technique: Preliminary result. Foot Ankle Surg. 2018 Aug;24(4):320-325. doi: 10.1016/j.fas.2017.03.002. Epub 2017 Mar 22. PMID 29409246
- [Background] Rigby RB, Cottom JM. A comparison of the "All-Inside" arthroscopic Brostrom procedure with the traditional open modified Brostrom-Gould technique: A review of 62 patients. Foot Ankle Surg. 2019 Feb;25(1):31-36. doi: 10.1016/j.fas.2017.07.642. Epub 2018 Feb 9. PMID 29409264
- [Background] Parisien JS, Shereff MJ. The role of arthroscopy in the diagnosis and treatment of disorders of the ankle. Foot Ankle. 1981 Nov;2(3):144-9. doi: 10.1177/107110078100200304. No abstract available. PMID 7341388
- [Background] Drez D Jr, Guhl JF, Gollehon DL. Ankle arthroscopy: technique and indications. Foot Ankle. 1981 Nov;2(3):138-43. doi: 10.1177/107110078100200303. No abstract available. PMID 7341387
- [Background] Glazebrook MA, Ganapathy V, Bridge MA, Stone JW, Allard JP. Evidence-based indications for ankle arthroscopy. Arthroscopy. 2009 Dec;25(12):1478-90. doi: 10.1016/j.arthro.2009.05.001. PMID 19962076
- [Background] Kerr HL, Bayley E, Jackson R, Kothari P. The role of arthroscopy in the treatment of functional instability of the ankle. Foot Ankle Surg. 2013 Dec;19(4):273-5. doi: 10.1016/j.fas.2013.06.008. Epub 2013 Jul 15. PMID 24095237
- [Background] Epstein DM, Black BS, Sherman SL. Anterior ankle arthroscopy: indications, pitfalls, and complications. Foot Ankle Clin. 2015 Mar;20(1):41-57. doi: 10.1016/j.fcl.2014.10.001. Epub 2014 Dec 15. PMID 25726482
- [Background] Schafer D, Hintermann B. Arthroscopic assessment of the chronic unstable ankle joint. Knee Surg Sports Traumatol Arthrosc. 1996;4(1):48-52. doi: 10.1007/BF01565998. PMID 8819064
- [Background] Ferkel RD, Karzel RP, Del Pizzo W, Friedman MJ, Fischer SP. Arthroscopic treatment of anterolateral impingement of the ankle. Am J Sports Med. 1991 Sep-Oct;19(5):440-6. doi: 10.1177/036354659101900504. PMID 1962707
- [Background] Ogilvie-Harris DJ, Gilbart MK, Chorney K. Chronic pain following ankle sprains in athletes: the role of arthroscopic surgery. Arthroscopy. 1997 Oct;13(5):564-74. doi: 10.1016/s0749-8063(97)90181-x. PMID 9343643
- [Background] Cameron SE, Wilson W, St Pierre P. A prospective, randomized comparison of open vs arthroscopically assisted ACL reconstruction. Orthopedics. 1995 Mar;18(3):249-52. doi: 10.3928/0147-7447-19950301-06. PMID 7761314
- [Background] Noyes FR, Mangine RE, Barber S. Early knee motion after open and arthroscopic anterior cruciate ligament reconstruction. Am J Sports Med. 1987 Mar-Apr;15(2):149-60. doi: 10.1177/036354658701500210. PMID 3555129
- [Background] Hohmann E, Tetsworth K, Glatt V. Open versus arthroscopic surgical treatment for anterior shoulder dislocation: a comparative systematic review and meta-analysis over the past 20 years. J Shoulder Elbow Surg. 2017 Oct;26(10):1873-1880. doi: 10.1016/j.jse.2017.04.009. Epub 2017 Jul 5. PMID 28688936
- [Background] Pulavarti RS, Symes TH, Rangan A. Surgical interventions for anterior shoulder instability in adults. Cochrane Database Syst Rev. 2009 Oct 7;(4):CD005077. doi: 10.1002/14651858.CD005077.pub2. PMID 19821339
- [Background] Corella F, Del Cerro M, Ocampos M, Simon de Blas C, Larrainzar-Garijo R. Arthroscopic Scapholunate Ligament Reconstruction, Volar and Dorsal Reconstruction. Hand Clin. 2017 Nov;33(4):687-707. doi: 10.1016/j.hcl.2017.07.019. PMID 28991581
- [Background] Shenoy K, Dai AZ, Mahure SA, Kaplan DJ, Capogna B, Youm T. Arthroscopic Repair of Hip Labrum With Suture Anchors. Arthrosc Tech. 2017 Nov 13;6(6):e2143-e2149. doi: 10.1016/j.eats.2017.08.007. eCollection 2017 Dec. PMID 29349010
- [Background] Guelfi M, Zamperetti M, Pantalone A, Usuelli FG, Salini V, Oliva XM. Open and arthroscopic lateral ligament repair for treatment of chronic ankle instability: A systematic review. Foot Ankle Surg. 2018 Feb;24(1):11-18. doi: 10.1016/j.fas.2016.05.315. Epub 2016 May 12. PMID 29413768